CLINICAL TRIAL: NCT07135141
Title: Mazdutide as Adjuvant Therapy Following Sleeve Gastrectomy in Severe Obesity:A Multicenter, Randomized, Double-Blind, Placebo-Controlled Superiority Trial
Brief Title: Mazdutide as Adjuvant Therapy Following Sleeve Gastrectomy in Severe Obesity
Acronym: SMART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Vice president of hospital, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMART trial
Record Dates: First submitted 2025-08-12; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve gastrectomy plus mazdutide group (Experimental): Participants will receive weekly subcutaneous injections of mazdutide at 5th month post sleeve gastrectomy(starting at 2.0 mg, with stepwise dose escalation to a target maintenance dose of 6.0 mg and optional adaptive downgrade to 4.0 mg if necessary)
  Interventions: Drug: Sleeve gastrectomy plus early mazdutide initiation
- Sleeve gastrectomy plus mazdutide placebo group (Placebo Comparator): Participants will receive weekly subcutaneous injections of matched placebo at 5th month post sleeve gastrectomy
  Interventions: Drug: Sleeve gastrectomy followed with early mazdutide placebo initation

INTERVENTIONS:
Drug: Sleeve gastrectomy plus early mazdutide initiation — After sleeve gastrectomy is preformed, mazdutide injection (pre-filled auto-injector pen) is administered subcutaneously at the same time each week at 5th month post procedure. The treatment begins with a starting dose of 2.0 mg, followed by a titration schedule increasing by 2.0 mg every 4 weeks (2.0 mg → 4.0 mg). If well-tolerated, participants reached the target maintenance dose of 6.0 mg (4.0 mg → 6.0 mg)weekly for maintenance. The protocol permits adaptive dose downgrade to 4.0 mg weekly when clinically indicated, such as intolerance. The total intervention is maintained until 48 weeks post procedure.
  Arms: Sleeve gastrectomy plus mazdutide group
Drug: Sleeve gastrectomy followed with early mazdutide placebo initation — After sleeve gastrectomy is preformed, mazdutide placebo injection (pre-filled auto-injector pen) is administered subcutaneously at the same time each week at 5th month post procedure. The treatment begins with a starting dose of 2.0 mg placebo, followed by a titration schedule increasing by 2.0 mg every 4 weeks (2.0 mg → 4.0 mg). If well-tolerated, participants reached the target maintenance dose of 6.0 mg placebo(4.0 mg → 6.0 mg) weekly for maintenance. The protocol permits adaptive dose downgrade to 4.0 mg weekly when clinically indicated, such as intolerance. The total intervention is maintained until 48 weeks post procedure.
  Arms: Sleeve gastrectomy plus mazdutide placebo group

SUMMARY:
The SMART study is a 96-week, multicenter, randomized, double-blind, placebo-controlled superiority clinical trial. A total of 256 severe obesity patients are randomized 1:1 to either receive the bariatric surgery plus GCG/GLP-1 dual receptor agonist group (receiving sleeve gastrectomy followed by subcutaneous injections of mazdutide weekly, with stepwise dose escalation to a maintenance dose per protocol) or the bariatric surgery plus placebo group (receiving matched procedure plus placebo injections). The primary objective is to evaluate the potential enhancing weight reduction effects of the combination therapy with bariatric surgery and mazdutide measured by the percentage change of excess weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years (inclusive), male or female;
* BMI≥37.5 kg/m2, with or without obesity-related complications;
* Planned to take sleeve gastrectomy
* Understand the trial protocol, voluntarily sign the informed consent form (ICF), and agree to follow all study requirements and restrictions.

Exclusion Criteria:

* Previous gastrointestinal surgery such as stomach and duodenum, or weight loss and metabolic surgery;
* History of thyroid C-cell carcinoma, multiple endocrine neoplasia (MEN) 2A or 2B, or relevant family history;
* ALT > 3.0 × ULN (if NAFLD is diagnosed at screening and within 6 months prior to screening, ALT ≤ 5.0 × ULN can be enrolled), or AST > 3.0 ×ULN, or total bilirubin (TBIL) > 2 × ULN
* Estimated glomerular filtration rate eGFR < 45 mL/min/1.73 m2 using the CKD-EPI equation
* Chronic anemia：Hemoglobin < 110 g/L (males) or < 100 g/L (females)；
* Have the following 12-lead electrocardiogram (ECGs) abnormalities at screening(<50 beats/min or >100 beats/min), 2nd or 3rd degree atrioventricular block, long QT syndrome or QTcF > 450 ms (males), QTcF > 470 ms (females), left or right bundle branch block, pre-excitation syndrome, or other significant arrhythmia (except sinus arrhythmia);
* Acute hyperglycemic/hypoglycemic events within 1 year, including:

diabetic ketoacidosis (DKA), hyperosmolar hyperglycemic state (HHS), and hypoglycemic coma, etc;

* Participants with previous severe myocardial infarction, stroke, acute and chronic heart failure, cardiac procedure such as percutaneous coronary intervention, coronary artery bypass grafting, or are not suitable for participation in this study after the investigator's assessment;
* Previous or confirmed mental illness at screening/randomization phase[Previous moderate to severe depressionPHQ questionnaire (Depression Screening Scale) ≥ 15 points, C-SSRS questionnaire (Columbia Suicide Severity Scale) category 4 or 5 at screening or randomization, or "Yes" in suicidal behavior or suicidal ideation];
* Previous specific infectious diseases, incl. acquired immunodeficiency syndrome, viral hepatitis B, viral hepatitis C, etc;
* End-stage disease with an expected survival of less than 5 years or previous/current malignancy;
* Use of GLP-1 receptor (GLP-1R) agonists or GLP-1R/GCGR agonists or GIPR/GLP-1R agonists or GIPR/GLP-1R/GCGR agonists within three months prior to screening;
* History of alcohol or drug abuse at screening;
* History of specific drugs use beyond 2 times, incl. moderate anticholinergics, antiparkinsonians, antiepileptic drugs, antipsychotics, benzodiazepines and sedatives, morphine and narcotic analgesics, stimulant drugs, medical marijuana, marijuana, and cannabidiol, etc.;
* Pregnant or lactating females, males or females of childbearing potential who are not willing to use contraception throughout the study and for 8 weeks after the end of the study;
* Having participated in other clinical investigators who have a conflict of interest with this study;
* The investigator suspects that the participant may be allergic to ingredients in the study drug or drugs of the same class;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
the rate of excess weight loss(EWL%) compared to baseline | At 48th week post procedure
  EWL%=[preoperative weight-post operative weight]/[preoperative weight -ideal body weight]x100%, ideal weight=height²(m²)x25kg/m²

SECONDARY OUTCOMES:
Assessing the change in BMI(kilogram/square meter, kg/m²） classification compared to baseline(Based on the BMI classification in Chinese adiposity diagnosis and treatment guideline 2024) | At 48th week post procedure
  BMI classification in China: BMI 18.5-24 kg/m² healthy; 24<BMI<28 kg/m² overweight, 28<BMI<32.5 kg/m² mild obesity, 32.5<BMI<37.5 kg/m² moderately obese, BMI>37.5 kg/m² severe or extremely severe obesity
Assessing the rate of total body weight loss(TBWL%) compared to baseline | At 48th week post procedure
  Total body weight loss (TBWL) is the pre-op weight minus the post op body weight
Assessing the change of waist circumference(centimeter, cm) compared to baseline | at 48th week post procedure
  waist circumference is measured with centimeter(cm)
Assessing the change of hip circumference(centimeter, cm) compared to baseline | At 48th week post procedure
  Hip circumference is measured with centimeter(cm).
Assessing the change of blood pressure(incl. systolic blood pressure and diastolic blood pressure) compared to baseline（Hydrargyrum, mmHg） | At 48th week post procedure
  Blood pressure is measured with mmHg.
Assessing the percentage change（%） of body fat or fat-free mass compared to baseline | At 48th week post procedure
  Body fat or fat-free mass is measured by dual energy X-ray absorptiometry(DEXA)
Assessing the percentage change（%） of liver fat content or pancreatic fat content compared to baseline | At 48th week post procedure
  Liver fat content or pancreatic fat content is measured with Magnetic resonance imaging-derived proton density fat fraction(MRI-PDFF)
Assessing the percentage change(%) of triglyceride(TG), low-density lipoprotein cholesterol(LDL-C),total cholesterol(TC) or high-density lipoprotein cholesterol(HDL-C) compared to baseline | At 48th week post procedure
  TG(millimoles per liter, mmol/L) , LDL-C(millimoles per liter, mmol/L) ,TC(millimoles per liter, mmol/L) or HDL-C(millimoles per liter, mmol/L) is tested in the lab of study sites with local standards according to Chinese Guidelines for Lipid Management
Assessing the change of aspartate transaminase(AST) or alanine aminotransferase(ALT) compared to baseline | At 48th week post procedure
Assessing the change(%) of serum uric acid compared to baseline | At 48th week post procedure
  serum uric acid(micromoles per liter, µmol/L) is tested in the lab of study sites according to Chinese National Standards
Assessing the change of nutrition status (incl. albumin, victamin B12, folic acid or serum iron and so forth) compared to baseline | At 48th week post procedure
  Albumin(gram per liter, g/L), folic acid(nanomoles per liter,nmol/L), Victamin B12(picomole per liter, pmol/L), serum iron(milligrams per liter, mg/L) is tested in the lab of study sites according to Chinese National Standards
Assessing the change of body weight related life quality(IWQOL-Lite) , upper GI symptom scale(GERDQ) or overall life quality scale(SF-36) compared to baseline | At 48th week post procedure
  IWQOL-Lite Score ranges among 31-105, the higher the score, the poorer the quality of life; When GerdQ score ≥8 points, it means the risk of gastroesophageal reflux is high; SF-36 score includes 8 dimensions, and the total score equals mean transformed scores of 8 dimensions, the higher the score, the higher the quality of life, transformed score of each dimension=［（actual score-the lowest possible score）/general average possible score］×100
Assessing the rate(%) of procedure-related or drug-related complications, re-admission, or major cardiovascular adverse events | At 48th week post procedure
  Procedure-related complications include gastroesophageal reflux disease, malnutrition and so on; Drug-related complications include nausea, vomiting, diarrhea and so on
Assessing the rate(%) of body weight regain among participants | At 96th week post procedure
  'Body weight rebounded over 15% compared to nadir weight' is referred to as weight regain

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Peking University People's Unviersity, Beijing
  - The Third Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Jinan University(Guangzhou Overseas Chinese Hospital), Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Kunming First People's Hospital, Kunming
  - Nanjing Drum Tower Hospital, Nanjing
  - Huadong Hospital affiliated to Fudan University, Shanghai
  - Shanghai Sixth People's Hospital to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjing
  - Zhongnan Hospital of Wuhan University, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR